CLINICAL TRIAL: NCT01739894
Title: Feasibility Study of Intraperitoneal Paclitaxel With Oxaliplatin and Capecitabine in Patients With Advanced Gastric Cancer
Brief Title: Feasibility Study of Intraperitoneal Paclitaxel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Yong Wei Peng, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA01/12/12
Record Dates: First submitted 2012-10-15; First posted 2012-12-04 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: Advanced gastric cancer; unresectable gastric cancer; recurrent gastric cancer; with peritoneal metastasis; cancer cells on peritoneal cytology
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IP Paclitaxel (Experimental): Paclitaxel will be administered intraperitoneally at 40mg/m2 on Days 1 and 8 in a 21-day cycle in patients receiving intravenous oxaliplatin 100mg/m2 on Day 1 and capecitabine 1000mg/m2 twice daily on Days 1-14.
  Interventions: Drug: IP Paclitaxel

INTERVENTIONS:
Drug: IP Paclitaxel — Each treatment cycle will consist of 21 days, with 14 days on treatment and 7 days off-treatment. Oxaliplatin will be administered intravenously (on Day 1 of each cycle). Paclitaxel will be administered intra-abdominally on Day 1 and Day 8 of each cycle. In particular, a needle will be inserted into the intraperitoneal injection port for normal saline to be injected intra-abdominally over one hour, followed by paclitaxel chemotherapy over a further one hour. Capecitabine will be taken by mouth from Day 1 to 14 of each cycle.

SUMMARY:
This is a single arm phase 2 trial evaluating the efficacy and tolerability of intraperitoneal paclitaxel with oxaliplatin and capecitabine in advanced gastric cancer patients with peritoneal metastasis and/or cancer cells on peritoneal cytology. Twenty patients will be recruited into the study for an estimated period of two years. Paclitaxel will be administered intraperitoneally at 40mg/m2 on Day 1 and 8 in patients receiving standard intravenous oxaliplatin 130mg/m2 on Day 1 and capecitabine 1000mg/m2 on day 1-14. The study hypothesizes that the addition of intraperitoneal paclitaxel with chemotherapy will improve treatment efficacy.

DETAILED DESCRIPTION:
The median survival of patients with unresectable gastric cancer treated with systemic chemotherapy is about 12 months. In patients with histologically proven unresectable or recurrent gastric cancer limited to the peritoneum and/or cancer cells in peritoneal cytology, the combination of i.p. paclitaxel with systemic chemotherapy reported a median survival time of 23.6 months. The peritoneal cytology turned negative for 86% of patients. In an updated report, gastrectomy was performed on 52 patients after disappearance or obvious shrinkage of peritoneal metastasis. In this cohort, the median survival time (MST) was 34.9 months. A phase III trial (PHOENIX-GC trial (Phase III study of S-1 plus intravenous and intraperitoneal paclitaxel versus S-1 plus cisplatin for gastric cancer with peritoneal metastasis )) comparing intraperitoneal(IP) regimen with systemic chemotherapy versus systemic therapy alone is currently opened for recruitment in Japan.

The multidisciplinary treatment combining IP-containing chemotherapy and surgery was found to be safe and effective for gastric cancer patients with peritoneal metastasis. A phase I study combining i.p. paclitaxel with oxaliplatin and S-1, found no dose limiting toxicity in all dose levels. Grade 3 neutropenia was observed in one patient at recommended phase 2 dose (RP2D) of i.p. paclitaxel of 40 mg/m2. In addition, grade 2 non-hematological toxicities observed were anorexia (n=6/12), fatigue (n=4/12) and nausea (n=2/12).

Both S-1 and capecitabine are orally available fluoropyrimidine. When combined with oxaliplatin, both S-1 and capecitabine were found to be equally active and well tolerated in advanced gastric cancer patients. As S-1 is not yet widely available worldwide, the combination of capecitabine and a platinum chemotherapy is still one of the most commonly adopted chemotherapy regimen for patients with advanced gastric cancer. In this study, we intend to assess the efficacy and feasibility of combining weekly i.p. paclitaxel with oxaliplatin and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven unresectable or recurrent adenocarcinoma of stomach and gastroesophageal junction
* Patients without prior systemic treatment. Patients who completed postoperative adjuvant chemotherapy (and radiotherapy) more than 180 days before may be enrolled
* Peritoneal metastasis and/or cancer cells on peritoneal cytology
* Age >21 years
* Eastern Cooperative Oncology Group performance status 0-2
* Adequate bone marrow function (neutrophil count >1500/mm3, hemoglobin >8.0 g/dl and platelet count >100 000/mm3)
* Adequate liver function (bilirubin, AST (aspartate aminotransferase)/ALT (alanine aminotransferase) within upper limit of normal)
* Adequate renal function (serum creatinine within the upper limit of normal)
* Expected survival >3 months
* Able to take orally
* Able to understand and the willingness to sign a written informed consent document
* The effects of proposed regimen on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antitumor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Metastasis to distant organ sites (such as the liver, lungs or bone)
* When trastuzumab is considered for palliative chemotherapy
* Known allergy to taxane, fluoropyrimidine or oxaliplatin
* Previous malignancy other than gastric cancer diagnosed in the last 5 years except for basal cell carcinoma of skin or preinvasive cancer of cervix
* Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients)
* Significant disease or conditions which, in the investigator's opinion, would exclude patient from the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating female

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-11 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) rate | 1 year
  The primary end point is 1-year survival because most patients may not have measurable disease, hence response rate and progression free survival are less easy to assess.

SECONDARY OUTCOMES:
Number of participants with adverse events | 3-weekly
  Toxicity will be monitored 3-weekly and graded according to the National Cancer Institute -Common Terminology Criteria for Adverse Events version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Ishigami H, Kaisaki S, Yamaguchi H et al. Phase I study of weekly intraperitoneal paclitaxel combined with S-1 and oxaliplatin for gastric cancer with peritoneal metastasis. J Clin Oncol 30, 2012 (suppl 4; abstr 146)
- [Background] Kim GM, Jeung HC, Rha SY, Kim HS, Jung I, Nam BH, Lee KH, Chung HC. A randomized phase II trial of S-1-oxaliplatin versus capecitabine-oxaliplatin in advanced gastric cancer. Eur J Cancer. 2012 Mar;48(4):518-26. doi: 10.1016/j.ejca.2011.12.017. Epub 2012 Jan 12. PMID 22243774
- [Background] Ishigami H, Kitayama J, Kaisaki S, Hidemura A, Kato M, Otani K, Kamei T, Soma D, Miyato H, Yamashita H, Nagawa H. Phase II study of weekly intravenous and intraperitoneal paclitaxel combined with S-1 for advanced gastric cancer with peritoneal metastasis. Ann Oncol. 2010 Jan;21(1):67-70. doi: 10.1093/annonc/mdp260. Epub 2009 Jul 15. PMID 19605503
- [Derived] Chia DKA, Ang JJ, Sundar R, Kim G, Shabbir A, So JBY, Yong WP. ASO Author Reflections: Combination Intra-Peritoneal and Systemic Chemotherapy for Gastric Cancer with Peritoneal Metastases. Ann Surg Oncol. 2022 Dec;29(13):8606-8607. doi: 10.1245/s10434-022-12102-1. Epub 2022 Oct 3. No abstract available. PMID 36192514